CLINICAL TRIAL: NCT03544892
Title: The Effects of a Low Carbohydrate, Non-Ketogenic Diet Versus Standard Diabetes Diet on Glycemic Control in Type 1 Diabetes
Acronym: T1DLoCHO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the University; study will not continue.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 8840
Record Dates: First submitted 2018-05-07; First posted 2018-06-04 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Low carbohydrate diet
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Intervention Model Description: This study uses 33 week randomized, powered study design to measure glycemic control with a low carbohydrate dietary pattern versus standard of care diabetes medical nutrition therapy. Each arm is 12 weeks with an 8 week washout between arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Low carbohydrate diet (Experimental)
  Interventions: Other: Low carbohydrate diet
- Experimental: Standard of care diet (Active Comparator)
  Interventions: Other: Standard of care diet

INTERVENTIONS:
Other: Low carbohydrate diet — 60-80 g total carbohydrate per day
  Arms: Experimental: Low carbohydrate diet
Other: Standard of care diet — > 150 g total carbohydrate per day
  Arms: Experimental: Standard of care diet

SUMMARY:
This randomized, crossover nutrition intervention seeks to examine the effects of a non-ketogenic low carbohydrate (CHO) diet (60-80g per day) on glycemic control, lipids, and markers on inflammation in individuals with Type 1 Diabetes (T1D). This study will be used to inform clinical practice, especially in teaching medical nutrition therapy to new-onset diabetes patients and those struggling with glycemic control and hyperlipidemia. At this time, no evidenced-based universal recommendations from randomized controlled trials exist to support low carbohydrate dietary patterns as a front-line approach in individuals with T1D. The investigators hypothesize a diet consisting of 60-80 g carbohydrate diet will result in greater improvement in glycemic control compared to a 50% carbohydrate diet in patients with Type 1 diabetes over 12 weeks in the outpatient setting.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1D) is marked by total insulin dependence with challenges regarding glycemic control and concomitant sequela. While standard of care medical nutrition therapy for this disease centers on matching carbohydrate to insulin at meals, recent literature and clinical reports have shown superior glycemic control and cardiovascular measures with lower carbohydrate dietary patterns (<130g/day) as compared to the standard American MyPlate (50% total calories as carbohydrate) approach. Diabetes management has evolved tremendously in the last twenty years with the development of sophisticated insulin pumps and continuous glucose monitors; but, glycemic control is still dependent on quantification of carbohydrate, imperfect in the real-world setting. Due to inherent error in carbohydrate counting, the investigators propose that less carbohydrate will produce better glycemic control by minimizing error and subsequent variation in individuals with type 1 diabetes.

There has long been a movement in the medical community to prescribe low carbohydrate diets under the premise of "less carbohydrate, less insulin, less glycemic variation". This strategy centers on "the law of small numbers", a calculus principle describing magnitude of variation in the output (glycemic variation) as the function of input size (CHO + insulin). Carbohydrate counting tends to result in ~50% error while there is ~30% variation in insulin action, making exactitude impossible. However, low CHO diets tend to provide >40% energy from fat due to the macronutrient distribution. With innate risk of cardiovascular disease in T1D, standard of care has supported restriction of total fat consumption, especially saturated fat, in effort to control cholesterol. While the American Diabetes Association recognizes that dietary fat is a controversial and complex issue, eliminating trans-fats is the only consensus point across the field. To date, most low CHO diet studies in both T1D and Type 2 Diabetes (T2D) have not shown adverse effects on lipids and tend to show decreases in triglycerides and either no change or increases in HDL, LDL, and total cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Type 1 diabetes for > 1 year confirmed by physician diagnosis
* HbA1c >5.9% and <10%;
* Confirmation of minimum three blood glucose tests per day (meter download or chart record)
* Use of continuous subcutaneous insulin infusion therapy (CSII) or multiple daily injection (MDI) intensive insulin therapy
* No change in insulin therapy type (CSII or MDI) in last 2 months or longer
* Willingness to count carbohydrate and use bolus calculator on insulin pump during the intervention periods
* Willingness to wear a 7 day CGM at three different time points during the study

Exclusion Criteria:

* Females of childbearing potential who are pregnant or intend to become pregnant, are exclusively breastfeeding, or who are not using adequate contraceptive methods
* Use of corticosteroids during or within 30 days prior to the intervention periods
* Macroalbuminuria
* Active proliferative retinopathy combined with an HbA1c ≥ 9%
* Known or suspected alcohol or drug abuse
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the patient unsuitable for study participation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Time in Range | 5 days of worn CGM during each intervention
  Difference in time spent with glucose values between 70-180 mg/dL assessed by continuous glucose monitoring (CGM)

SECONDARY OUTCOMES:
Mean Glucose | Baseline to 12 weeks (1 week worn CGM data)
  Difference in mean glucose values assessed by CGM
Standard deviation of glucose | Baseline to 12 weeks (1 week worn CGM data)
  Difference in standard deviation of glucose values assessed by CGM
Mean amplitude of glycemic excursions | Baseline to 12 weeks (1 week worn CGM data)
  Difference in mean amplitude of glycemic excursions assessed by CGM
Time in hypoglycemia | Baseline to 12 weeks (1 week worn CGM data)
  Difference in time spent with glucose values <70 mg/dL; between 55-70 mg/dL; and <55 mg/dL
Time in hyperglycemia | Baseline to 12 weeks (1 week worn CGM data)
  Difference in time spent with glucose values >180 mg/dL
Change in HbA1c | Baseline to 12 weeks
  Difference in change in hemoglobin A1c
Coefficient of Variation | Baseline to 12 weeks (1 week worn CGM data)
  Estimate of glucose variability calculated by dividing the standard deviation by average glucose
Severe hypoglycemia | Baseline to 12 weeks
  Difference in number of severe hypoglycemia episodes (glucagon or IV dextrose administration)
Total daily insulin dose | Baseline to 12 weeks
  Difference in total daily insulin dose
Total daily basal insulin 24 hour | Baseline to 12 weeks
  Difference in total daily basal insulin in 24 hours
Total daily bolus insulin 24 hour | Baseline to 12 weeks
  Difference in total daily bolus insulin in 24 hours
Body weight | Baseline to 12 weeks
  Change in body weight
Body Mass Index (BMI) | Baseline to 12 weeks
  Change in BMI
Systolic Blood Pressure (mm Hg) | Baseline to 12 weeks
  Change in systolic BP
Diastolic Blood Pressure (mm Hg) | Baseline to 12 weeks
  Change in diastolic BP
Pulse, per minute | Baseline to 12 weeks
  Change in pulse
Energy Intake (kcal/day) | Baseline to 12 weeks
  Change in energy intake
Daily carbohydrate intake (total carbohydrate, g/day) | Baseline to 12 weeks
  Change in carbohydrate intake
Percent energy intake as Carbohydrate | Baseline to 12 weeks
  Change in % carbohydrate intake
Daily protein intake (total protein, g/day) and Daily fat intake (total fat, g/day) | Baseline to 12 weeks
  Change in protein intake
Fat quality intake (% total fat as monounsaturated, polyunsaturated, saturated, omega-3) | Baseline to 12 weeks
  Change in fat quality
Standard Lipid Panel | Baseline to 12 weeks
  Change in (Total cholesterol, HDL cholesterol, LDL cholesterol-calculated, triglycerides; mg/dL)
LDL-P (nmol/L) | Baseline to 12 weeks
  Change in LDL-P
HDL-P (umol/L) | Baseline to 12 weeks
  Change in HDL-P
VLDL-P | Baseline to 12 weeks
  Change in VLDL-P (nmol/L)
LDL size | Baseline to 12 weeks
  Change in LDL size (nm)
HDL size | Baseline to 12 weeks
  Change in HDL size (nm)
VLDL size | Baseline to 12 weeks
  Change in VLDL size (nm)
High-sensitive C-reactive protein (hs-CRP) | Baseline to 12 weeks
  Change in hs-CRP
Plasma lipopolysaccharide | Baseline to 12 weeks
  Surrogate marker for inflammation
Serum Ketones (beta-hydroxybutyrate) | Baseline to 12 weeks
  beta-hydroxybutyrate (mmol/L)
Type 1 Diabetes Nutrition Knowledge Survey | Baseline to Week 33 (end of study)
  Validated nutrition knowledge survey (nutrition label reading, carbohydrate counting)
Diet Quality | Baseline to 12 weeks
  Minerals, Vitamins, Dietary Fiber amounts compared to DRIs for age, ascertained by 3 day 24 hour food logs

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Crowder, RDN, CNSC, LD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Harold Hamm Diabetes Center, Tulsa, Oklahoma, United States